CLINICAL TRIAL: NCT03633760
Title: A Different Level of Single-dose and Multiple-dose Study to Evaluate the Pharmacokinetics of Bilastine in a Chinese Population
Brief Title: Different Level of Single-dose and Multiple-dose Bilastine PK Study in Chinese Population
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.Menarini Asia-Pacific Holdings Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: INCN/12/Bil-PK/004
Record Dates: First submitted 2018-08-03; First posted 2018-08-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — bilastine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilastine 40mg single dose (Experimental): 12 eligible subjects will be allocated to this arm and receive a single dose of 40 mg of bilastine
  Interventions: Drug: Bilastine 40mg single dose
- Bilastine 20mg multiple dose (Experimental): 12 eligible subjects will be allocated to this arm and receive a single dose of bilastine 20 mg on Day 1 and six doses of bilastine 20 mg from Day 4 to Day 9
  Interventions: Drug: Bilastine 20mg single-dose followed by multiple-dose

INTERVENTIONS:
Drug: Bilastine 40mg single dose — Single-dose only cohort treatment duration is 1 day. After the screening period, eligible subjects will be allocated to receive a single dose of 40 mg of bilastine
  Arms: Bilastine 40mg single dose
Drug: Bilastine 20mg single-dose followed by multiple-dose — Single-dose followed by multiple-dose cohort treatment duration of this cohort is 9 days. Subjects will receive a single dose of bilastine 20 mg on the morning of Day 1; and six doses of bilastine 20 mg in the morning from Day 4 to Day 9.
  Arms: Bilastine 20mg multiple dose

SUMMARY:
This is a single-dose and multiple-dose, open-label, single-centre pharmacokinetic (PK) study which will be conducted in Phase I Clinical Trial Centre, Chinese University of Hong Kong, to evaluate pharmacokinetics (PK) of different levels of single-dose and multiple-dose of bilastine in healthy Chinese subjects.

DETAILED DESCRIPTION:
This is a single-dose and multiple-dose, open-label, single-centre pharmacokinetic (PK) study, to evaluate pharmacokinetics (PK) of different levels of single-dose and multiple-dose of bilastine in healthy Chinese subjects. Total 24 subjects will be enrolled into the study and divided into 2 cohorts, 12 subjects in each cohort.

Single-dose only cohort treatment duration is 1 day and receive a single dose of 40 mg of bilastine then collect PK blood sample. Single-dose followed by multiple-dose cohort treatment duration of this cohort is 9 days. Subjects will receive a single dose of bilastine 20 mg on the morning of Day 1; and six doses of bilastine 20 mg in the morning from Day 4 to Day 9 and collect PK blood samples. The primary objective of the study is to determine the PK properties of orally administered bilastine in healthy Chinese population. The secondary objective of the study is to evaluate the safety and tolerability of bilastine administered as a single and multiple doses in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese males and females between 18 and 45 years of age (inclusive).
2. Having voluntarily given their informed consent to participate in the study after receiving information about the design, aims and potential risks that could result from the study and being informed that they could refuse to take part in or withdraw from the study at any time.
3. Body mass of no less than 50 kg. Body mass index: 19 to 24 kg/m2 (inclusive).
4. No clinically significant abnormal findings from the physical examination, vital signs check, electrocardiogram (ECG), medical history, or clinical laboratory results during screening and pre-dosing of Day 1.
5. A negative screen for HIV and hepatitis B.
6. A negative urine or breathalyzer screen for alcohol and negative urine screen for drugs of abuse.
7. Are non-tobacco / nicotine users (within 3 months prior to screening visit).
8. A negative serum pregnancy test for female subjects.
9. Subjects who are willing to comply with the contraception restrictions for this study:

   1. True abstinence.
   2. Barrier methods with spermicidal use. The use of barrier contraceptives should always be supplemented with the use of a spermicide, where available.
   3. Intrauterine devices: intrauterine device with the use of condom or spermicide.
   4. Sterilization of male subjects (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).

Exclusion Criteria:

1. History of clinically significant gastrointestinal, renal, hepatic, neurologic, haematological, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, jeopardises the safety of the subject or will impact the validity of the study results.
2. History of allergic or adverse response to antihistamine drugs.
3. Participated in a clinical trial within 90 days prior to screening.
4. Donated blood within 90 days prior to screening.
5. Donated plasma within 90 days prior to screening.
6. Abnormal diet or substantial changes in eating habits within 30 days prior to screening.
7. Used any prescription medication within 14 days prior to or during screening, especially any known P-glycoprotein transporter inhibitors agents (ketoconazole, erythromycin, ciclosporin, digoxin, etc.).
8. Used any prescription or any over-the-counter medication, herbal or traditional Chinese medication within 7 days prior to or during screening.
9. Intake of grapefruit or any other citrus fruit, fruit juice or cranberries within 72 hours prior to study drug administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (Cmax) | day1, day4 to day9
  observed maximum plasma concentration
Pharmacokinetic (tmax) | day1, day4 to day9
  time to reach Cmax
Pharmacokinetic (λz) | day1, day4 to day9
  terminal rate constant
Pharmacokinetic (t½) | day1, day4 to day9
  terminal half-life
Pharmacokinetic [AUC(0-24)] | day1
  area under the plasma concentration-time curve from zero to 24 hours after study drug administration
Pharmacokinetic [AUC(0-last)] | day1
  from time zero to the time of last quantifiable concentration
Pharmacokinetic [AUC(0-inf)] | day1
  from time zero extrapolated to infinity
Pharmacokinetic (CL/F) | day1, day4 to day9
  apparent systemic clearance following oral dosing
Pharmacokinetic (Vz/F) | day1, day4 to day9
  apparent volume of distribution during terminal phase following oral dosing
Pharmacokinetic [AUC(0-inf)/D] | day1
  dose-normalized AUC(0-inf)
Pharmacokinetic (Cmax/D) | day1
  dose-normalized Cmax
Pharmacokinetic (Cavg) | day4 to day9
  average concentration over the study drug interval
Pharmacokinetic [AUC(0-tau)] | day4 to day9
  area under the plasma concentration-time curve during the dosing interval following multiple dosing
Pharmacokinetic (FI) | day4 to day9
  fluctuation index
Pharmacokinetic (LI) | day4 to day9
  linearity index
Pharmacokinetic [RAUC(0-tau)] | day4 to day9
  accumulation ratio for AUC(0-tau)
Pharmacokinetic (RCmax) | day4 to day9
  accumulation for Cmax

SECONDARY OUTCOMES:
Adverse events | day1 to day16
  Safety will be evaluated with summary of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Luk, Professor, Principal Investigator — Phase I Clinical Trial Centre, Chinese University of Hong Kong
Locations (1):
- Phase I Clinical Trial Centre, Chinese University of Hong Kong, Hong Kong, Hong Kong, China